CLINICAL TRIAL: NCT02263027
Title: Do Some Healthy Adults Consistently Have Systemic Reactions to Trivalent Inactivated Split Virus Influenza Vaccines?
Brief Title: Do Some Healthy Adults Consistently Have Systemic Reactions to Influenza Vaccines?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 14-0808
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-09

CONDITIONS: Influenza
Keywords: influenza vaccine; adult; safety; reactogenicity
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccine, then placebo (Experimental): 1 injection of trivalent inactivated influenza vaccine, 0.5mL/dose, as approved for use in Canada for season of enrolment followed by 1 injection of normal saline placebo, 0.5mL/dose, 28 days later
  Interventions: Biological: Vaccine
- Placebo, then vaccine (Experimental): 1 injection of normal saline placebo, 0.5mL/dose followed by 1 injection of trivalent inactivated influenza vaccine, 0.5mL/dose, as approved for use in Canada for season of enrolment, 28 days later
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — Licensed trivalent inactivated influenza vaccine
  Other Names: Trivalent inactivated influenza vaccine

SUMMARY:
This study will recruit 35 healthcare workers who had systemic reactions to influenza vaccine the last 2 times they were vaccinated, to ask whether influenza vaccine is indeed associated with systemic reactions in these workers.

DETAILED DESCRIPTION:
Randomized controlled trials of split virus vaccines in healthy adults have not been able to detect an increase in systemic adverse events compared to control vaccination. These trials do identify a non-trivial risk of systemic symptoms occurring in the week after both placebo and vaccine. There is a small population of healthcare workers who report consistent systemic symptoms after split virus vaccination which may occur because a small group of healthy adults have true physical reactions to components of the vaccine or excipients. If this is true, then alternatives - such as the use of subunit vaccines or live attenuated nasal spray vaccines - might be expected to be better tolerated by these people.

ELIGIBILITY:
Inclusion Criteria:

* Employed or volunteer in a healthcare facility or an ambulatory care setting providing healthcare
* By self report, have had 2 or more doses of trivalent inactivated influenza vaccine (TIIV) in the last 15 years, and after at least the last 2 vaccine doses have had the same systemic adverse event in the 7 days after vaccination, including: fever, chills, myalgia, arthralgia, fatigue, headache, or insomnia;
* Consent to the study, including two injections one month apart, with one being placebo and one a dose of TIIV;

Exclusion Criteria:

* Has a contraindication to TIIV (previous allergic reaction to a dose of vaccine, or Guillain Barre syndrome with onset within 6 weeks of vaccination);
* Has previously received a dose of TIIV for the current influenza season.
* Receipt of another vaccine, or initiation of new medication within 7 days of the study injection (participant may enter the study as long as the gap between other vaccine/initiation of new medication is >7 days);
* Moderate or severe acute illness or active infection or fever (temperature ≥37.8oC) on the day a dose of study medication due (participant may receive injection 48 hours after symptoms have resolved and body temperature has returned to normal without the use of antipyretics.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Systemic adverse event | 7 days after each injection
  Any systemic adverse event, self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Allison J McGeer, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada